CLINICAL TRIAL: NCT00881426
Title: Comparative, Randomized, Single-Dose, 2-way Crossover Bioavailability Study of Sandoz GmbH and Bristol-Myers Squibb (Cefzil) 500 mg Cefprozil Tablets In Healthy Adults Volunteers Under Fasting Conditions
Brief Title: To Demonstrate the Relative Bioavailability of Cefzil 500 mg Cefprozil Tablets Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sandoz (Industry)
Responsible Party: Eric Mittleberg, Ph.D, VP of Product Development, Sandoz Inc.
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AA17499
Record Dates: First submitted 2009-04-14; First posted 2009-04-15 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2009-04

CONDITIONS: Healthy
Keywords: Antibiotic
MeSH Terms: interventions — Cefprozil

ARMS (2):
- 1 (Experimental): Cefprozil 500 mg Tablets (Sandoz GmbH)
  Interventions: Drug: Cefprozil 500 mg Tablets (Sandoz GmbH)
- 2 (Active Comparator): Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb)
  Interventions: Drug: Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb)

INTERVENTIONS:
Drug: Cefprozil 500 mg Tablets (Sandoz GmbH)
  Arms: 1
Drug: Cefzil (Cefprozil) 500 mg Tablets (Bristol-Myers Squibb)
  Arms: 2

SUMMARY:
To demonstrate the relative bioavailability of Cefzil 500 mg Cefprozil tablets under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal finding on physical exam, medical history, or clinical laboratory results on screening.

Exclusion Criteria:

* Positive test results for HIV or hepatitis B or C.
* Treatment for drug or alcohol dependence.

Ages: 20 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-03; Primary Completion 2004-04 (Actual); Study Completion 2004-04 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on AUC and Cmax | 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Gaetano Morelli, M.D., Principal Investigator — MDS Pharma Services